CLINICAL TRIAL: NCT03900416
Title: Mindfulness-based Mobile Application to Reduce Rumination in Adolescents
Brief Title: Adolescent Mindfulness Mobile App Study (RCT)
Acronym: AMMASRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lawrence University (Other)
Responsible Party: Principal Investigator, Lori Hilt, Associate Professor of Psychology, Lawrence University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7_25_18_Hilt
Record Dates: First submitted 2019-03-22; First posted 2019-04-03 (Actual); Results first posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: Rumination; Depression; Anxiety; Self-Injurious Behavior
Keywords: Mindfulness; Mobile Intervention; Brief Intervention; Adolescence
MeSH Terms: conditions — Rumination Syndrome; Depression; Anxiety Disorders; Self-Injurious Behavior

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to the intervention group (i.e., mindfulness with ecological momentary assessment) or the control group (i.e., ecological momentary assessment only).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness App (Experimental): Guided mindfulness exercises will be delivered via mobile app for three weeks.
  Interventions: Behavioral: Mindfulness App
- Control condition (No Intervention): Participants will use app for assessment for three weeks, but no mindfulness exercises will be delivered.

INTERVENTIONS:
Behavioral: Mindfulness App — Mindfulness exercises will last 1-12 minutes. Each one asks participants to focus on something (e.g., breath, sounds, physical sensations) using guided instruction.
  Arms: Mindfulness App

SUMMARY:
Rumination involves focusing on negative emotions repeatedly and is a risk factor for developing depression, anxiety, and self-injury. These negative outcomes increase in adolescence. The main goal of this study is to examine whether a mobile application designed to reduce rumination works with adolescents. The mobile application involves mindfulness exercises. Mindfulness means nonjudgmentally and deliberately paying attention. Adolescents will be randomly assigned to either the mindfulness group or a control group who uses a mobile application without mindfulness exercises. Both groups will use the app three times per day for three weeks and we will follow up with participants for six months. The investigators hypothesize that the mindfulness group will experience a reduction in rumination and symptoms of depression, anxiety and self-injury. They also expect that the mindfulness group will find the mobile app to be more engaging and will continue to use it beyond the 3 weeks.

DETAILED DESCRIPTION:
Rumination, a perseverative cognitive process that involves dwelling on negative emotions, is a transdiagnostic risk factor for the development of depression, anxiety, and self-injurious behaviors. Thus, reducing the tendency to ruminate in adolescence, a time when many psychological disorders often first develop, has the potential for a large public health impact. This protocol involves testing the acceptability and efficacy of a newly developed mindfulness mobile application designed to reduce rumination.

Mindfulness involves paying attention to the present moment without judgement. If negative emotions arise, one notices them and how the body is feeling without becoming caught up in the emotion so that it can pass. In adult clinical studies, intensive mindfulness practice has been associated with successful treatment of psychopathology, including preventing the recurrence of depression, possibly through reducing rumination. Research with adolescents has suggested that a brief mindfulness exercise can interrupt the ruminative process. Thus, mindfulness appears to be a promising strategy to reduce the tendency to ruminate and prevent psychopathology.

A diverse sample of 150 high-ruminating 12-15 year-olds will be recruited from the community and randomly assigned to a 3-week mobile mindfulness intervention or an ecological momentary assessment (EMA)-only control condition. In both conditions, adolescents will be notified to use the mobile app three times per day to complete EMA questions. Based on mood ratings, participants in the mindfulness condition have a chance to receive a brief mindfulness exercise (i.e., 1-12 minutes long) at each use. At pre- and post-intervention and three follow-up periods (6 weeks,12 weeks, and 6 months), participants and their parents will report on adolescent anxiety and depression. Adolescents will also report on self-injurious thoughts and behaviors (SITBs), trait rumination, and mindfulness. During the intervention period, participants will report on state levels of rumination, mindfulness, and mood using the app. Participants will also report on their satisfaction with the app, while their optional continued use of the app will be monitored electronically for 6 months following the intervention period. The investigators will test intervention effects using multilevel modeling, examining the role of both state- and trait-level mediators. Based on preliminary pilot data, the investigators expect that the mindfulness intervention will reduce symptoms, and we anticipate this effect to be due to the mediating role of decreased rumination.

ELIGIBILITY:
Inclusion Criteria:

* adolescent between the ages of 12 and 15 years
* at least moderate levels of rumination (mean score of 2 or above on a 1-4 scale) on the two screening questions

Exclusion Criteria:

* serious physical or cognitive disability that prevents adolescent from using a mobile device, because that is the intervention delivery method
* inadequate English proficiency to complete questionnaires

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 152 (Actual)
Dates: Start 2019-06-17 (Actual); Primary Completion 2021-02-03 (Actual); Study Completion 2021-02-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori M Hilt, PhD, Principal Investigator — Lawrence University
Locations (1):
- Lawrence University, Appleton, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hilt LM, Swords CM, Webb CA. Randomized Controlled Trial of a Mindfulness Mobile Application for Ruminative Adolescents. J Clin Child Adolesc Psychol. 2025 Jan-Feb;54(1):99-112. doi: 10.1080/15374416.2022.2158840. Epub 2023 Jan 9. PMID 36622879
- [Derived] Webb CA, Swords CM, Lawrence HR, Hilt LM. Which adolescents are well-suited to app-based mindfulness training? A randomized clinical trial and data-driven approach for personalized recommendations. J Consult Clin Psychol. 2022 Sep;90(9):655-669. doi: 10.1037/ccp0000763. PMID 36279218

RESULTS

PARTICIPANT FLOW:
Period: Baseline
Arm/Group | Mindfulness App | Control Condition
Started | 72 | 80
Completed | 72 | 80
Not Completed | 0 | 0
Period: Post
Arm/Group | Mindfulness App | Control Condition
Started | 72 | 80
Completed | 72 | 80
Not Completed | 0 | 0
Period: Six Week Follow-up
Arm/Group | Mindfulness App | Control Condition
Started | 72 | 80
Completed | 70 | 80
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Twelve Week Follow-up
Arm/Group | Mindfulness App | Control Condition
Started | 70 | 80
Completed | 69 | 76
Not Completed | 1 | 4
Not completed — Lost to Follow-up | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Adverse Event | 1 | 1
Period: Six Month Follow-up
Arm/Group | Mindfulness App | Control Condition
Started | 69 | 76
Completed | 64 | 72
Not Completed | 5 | 4
Not completed — Lost to Follow-up | 4 | 3
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness App | Control Condition | Total
Number analyzed (Participants) | 72 | 80 | 152
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.78 (.93) | 13.66 (.86) | 13.71 (.89)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Sex as reported by parent
  Participants
    Female | 44 | 45 | 89
    Male | 28 | 35 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 7 | 16
  Not Hispanic or Latino | 63 | 73 | 136
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Categorical measure, data collected at baseline
  Participants
    Race: White | 55 | 70 | 125
    Race: Black; African American | 3 | 2 | 5
    Race: Asian; Asian American | 1 | 2 | 3
    Race: Native Hawaiian or Pacific Islander | 1 | 0 | 1
    Race: Native American | 0 | 0 | 0
    Race: Multi-racial | 11 | 5 | 16
    Race: Other | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 72 | 80 | 152
Children's Response Styles Questionnaire [Mean (Standard Deviation); unit: units on a scale] — trait rumination (range = 0-39 with higher scores indicating more rumination)
  units on a scale | 33.47 (9.64) | 30.73 (9.05) | 32.03 (9.40)
Children's Depression Inventory [Mean (Standard Deviation); unit: units on a scale] — self-reported depressive symptoms (range = 0-54 with higher scores indicating more symptoms)
  units on a scale | 13.4 (8.77) | 12.04 (7.72) | 12.68 (8.23)
Multidimensional Anxiety Scale for Children [Mean (Standard Deviation); unit: units on a scale] — self-reported anxiety symptoms (range = 0-117 with higher scores indicating more anxiety)
  units on a scale | 53.47 (16.51) | 50.84 (17.35) | 52.09 (16.95)
Self-injurious Thoughts and Behaviors Questionnaire [Count of Participants; unit: Participants] — Self-reported lifetime engagement in nonsuicidal self-injury
  Participants | 11 | 11 | 22
Pediatric Symptom Checklist Internalizing Scale [Mean (Standard Deviation); unit: units on a scale] — parent-reported internalizing symptoms (range = 0-10 with higher scores indicating more internalizing symptoms)
  units on a scale | 3.64 (2.38) | 3.88 (2.45) | 3.76 (2.411)
Five Facet Mindfulness Questionnaire Observing Subscale [Mean (Standard Deviation); unit: units on a scale] — trait mindfulness observing (range = 8-40 with higher scores indicating greater mindfulness)
  units on a scale | 22.28 (6.23) | 21.38 (6.2) | 21.80 (6.206)
Five Facet Mindfulness Questionnaire Describing Subscale [Mean (Standard Deviation); unit: units on a scale] — trait mindfulness describing (range = 8-40 with higher scores indicating greater mindfulness)
  units on a scale | 24.26 (5.75) | 24.69 (5.75) | 24.49 (5.74)
Five Facet Mindfulness Questionnaire Awareness Subscale [Mean (Standard Deviation); unit: units on a scale] — trait mindfulness acting with awareness (range = 8-40 with higher scores indicating greater mindfulness)
  units on a scale | 25.03 (6.23) | 26.17 (5.84) | 25.63 (6.04)
Five Facet Mindfulness Questionnaire Nonjudging Subscale [Mean (Standard Deviation); unit: units on a scale] — trait mindfulness non-judging of inner experience (range = 8-40 with higher scores indicating greater mindfulness)
  units on a scale | 25.56 (7.46) | 27.49 (7.58) | 26.57 (7.561)
Five Facet Mindfulness Questionnaire Nonreactivity Subscale [Mean (Standard Deviation); unit: units on a scale] — trait mindfulness non-reactivity to inner experience (range = 7-35 with higher scores indicating greater mindfulness)
  units on a scale | 19.58 (4.58) | 19.44 (3.99) | 19.51 (4.268)

OUTCOME MEASURES:

1. Primary Outcome: Children's Response Styles Questionnaire
Description: trait rumination (range = 0-39 with higher scores indicating more rumination)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 72 | 80
score on a scale | 33.47 (9.64) | 30.73 (9.05)

2. Primary Outcome: Children's Response Styles Questionnaire
Description: trait rumination (range = 0-39 with higher scores indicating more rumination)
Time Frame: 3 weeks (i.e., immediately post-intervention)
Population: Number analyzed determined by number of adolescents that completed the questionnaire.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 71 | 79
score on a scale | 29.48 (9.89) | 30.76 (10.12)

3. Primary Outcome: Children's Response Styles Questionnaire
Description: trait rumination (range = 0-39 with higher scores indicating more rumination)
Time Frame: 6 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 66 | 76
score on a scale | 27.71 (9.46) | 29.17 (10.64)

4. Primary Outcome: Children's Response Styles Questionnaire
Description: trait rumination (range = 0-39 with higher scores indicating more rumination)
Time Frame: 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 64 | 74
score on a scale | 29.27 (10.22) | 28.45 (9.8)

5. Primary Outcome: Children's Response Styles Questionnaire
Description: trait rumination (range = 0-39 with higher scores indicating more rumination)
Time Frame: 6 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 63 | 71
score on a scale | 29.4 (10.79) | 29.77 (10.05)

6. Primary Outcome: Children's Depression Inventory
Description: self-reported depressive symptoms (range = 0-54 with higher scores indicating more symptoms)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 72 | 80
score on a scale | 13.4 (8.77) | 12.04 (7.72)

7. Primary Outcome: Children's Depression Inventory
Description: self-reported depressive symptoms (range = 0-54 with higher scores indicating more symptoms)
Time Frame: 3 weeks (immediately post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 71 | 79
score on a scale | 11.52 (9.54) | 12.22 (8.57)

8. Primary Outcome: Children's Depression Inventory
Description: self-reported depressive symptoms (range = 0-54 with higher scores indicating more symptoms)
Time Frame: 6 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 66 | 76
score on a scale | 10.68 (9.04) | 10.82 (8.23)

9. Primary Outcome: Children's Depression Inventory
Description: self-reported depressive symptoms (range = 0-54 with higher scores indicating more symptoms)
Time Frame: 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 64 | 74
score on a scale | 9.33 (7.97) | 10.54 (8.57)

10. Primary Outcome: Children's Depression Inventory
Description: self-reported depressive symptoms (range = 0-54 with higher scores indicating more symptoms)
Time Frame: 6 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 63 | 71
score on a scale | 8.84 (8.02) | 10.42 (8.97)

11. Primary Outcome: Multidimensional Anxiety Scale for Children
Description: self-reported anxiety symptoms (range = 0-117 with higher scores indicating more anxiety)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 72 | 80
score on a scale | 53.47 (16.51) | 50.84 (17.35)

12. Primary Outcome: Multidimensional Anxiety Scale for Children
Description: self-reported anxiety symptoms (range = 0-117 with higher scores indicating more anxiety)
Time Frame: 3 weeks (i.e., immediately post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 71 | 79
score on a scale | 50.94 (16.82) | 52.37 (17.64)

13. Primary Outcome: Multidimensional Anxiety Scale for Children
Description: self-reported anxiety symptoms (range = 0-117 with higher scores indicating more anxiety)
Time Frame: 6 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 66 | 76
score on a scale | 51.00 (16.52) | 49.88 (19.25)

14. Primary Outcome: Multidimensional Anxiety Scale for Children
Description: self-reported anxiety symptoms (range = 0-117 with higher scores indicating more anxiety)
Time Frame: 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 64 | 74
score on a scale | 50.34 (18.18) | 49.82 (19.11)

15. Primary Outcome: Multidimensional Anxiety Scale for Children
Description: self-reported anxiety symptoms (range = 0-117 with higher scores indicating more anxiety)
Time Frame: 6 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 63 | 71
score on a scale | 49.29 (16.74) | 49.56 (20.58)

16. Primary Outcome: Self-injurious Thoughts and Behaviors Questionnaire
Description: percent of participants engaged in self-injury over the past year
Time Frame: baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 72 | 80
Participants | 7 | 7

17. Primary Outcome: Self-injurious Thoughts and Behaviors Questionnaire
Description: percent of participants that engaged in self-injury over the past 3 weeks
Time Frame: 3 weeks (i.e., immediately post-intervention)
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 71 | 79
Participants | 1 | 2

18. Primary Outcome: Self-injurious Thoughts and Behaviors Questionnaire
Description: percent of participants that engaged in self-injury over the past 6 weeks
Time Frame: 6 weeks post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 66 | 76
Participants | 3 | 3

19. Primary Outcome: Self-injurious Thoughts and Behaviors Questionnaire
Description: percent of time engaged in self-injury over the past 6 weeks
Time Frame: 12 weeks post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 64 | 74
Participants | 2 | 1

20. Primary Outcome: Self-injurious Thoughts and Behaviors Questionnaire
Description: percent of time engaged in self-injury over the past 3 months
Time Frame: 6 months post intervention
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 63 | 71
Participants | 3 | 2

21. Primary Outcome: Pediatric Symptom Checklist Internalizing Scale
Description: parent-reported internalizing symptoms (range = 0-10 with higher scores indicating more internalizing symptoms)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 72 | 80
score on a scale | 3.64 (2.38) | 3.88 (2.45)

22. Primary Outcome: Pediatric Symptom Checklist Internalizing Scale
Description: parent-reported internalizing symptoms (range = 0-10 with higher scores indicating more internalizing symptoms)
Time Frame: 3 weeks (i.e., immediately post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 71 | 79
score on a scale | 2.49 (2.21) | 2.46 (1.99)

23. Primary Outcome: Pediatric Symptom Checklist Internalizing Scale
Description: parent-reported internalizing symptoms (range = 0-10 with higher scores indicating more internalizing symptoms)
Time Frame: 6 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 68 | 75
score on a scale | 2.38 (2.05) | 2.41 (2.09)

24. Primary Outcome: Pediatric Symptom Checklist Internalizing Scale
Description: parent-reported internalizing symptoms (range = 0-10 with higher scores indicating more internalizing symptoms)
Time Frame: 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 66 | 74
score on a scale | 2.49 (2.14) | 2.35 (2.14)

25. Primary Outcome: Pediatric Symptom Checklist Internalizing Scale
Description: parent-reported internalizing symptoms (range = 0-10 with higher scores indicating more internalizing symptoms)
Time Frame: 6 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 63 | 72
score on a scale | 2.38 (1.96) | 2.68 (2.26)

26. Primary Outcome: State Rumination
Description: average state rumination during intervention period rated on a visual analog scale (range = 0-100 with higher scores indicating more rumination)
Time Frame: 3 weeks (i.e., immediately post-intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 72 | 80
units on a scale
  Emotion-Focused Rumination | 41.88 (20.44) | 42.53 (20.17)
  Problem-Focused Rumination | 34.80 (18.47) | 37.58 (18.69)

27. Primary Outcome: State Mood
Description: average sadness and anxiety during intervention period rated on visual analog scales (range = 0-100 with higher scores indicating more rumination)
Time Frame: 3 weeks (i.e., immediately post-intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 72 | 80
units on a scale
  Anxiety | 36.62 (19.35) | 39.08 (20.05)
  Sadness | 25.00 (17.72) | 25.02 (14.10)

28. Primary Outcome: Daily App Use
Description: Daily app use was determined by how many complete app uses were logged during the three-week intervention period.
Time Frame: 3 weeks (i.e., immediately post-intervention)
Measure: Mean (Standard Deviation); unit: App uses
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 72 | 80
App uses | 51.72 (16.37) | 54.26 (15.26)

29. Primary Outcome: Continued Use
Description: Number of times app was used after the 3 week intervention period
Time Frame: 6 months post intervention
Measure: Mean (Standard Deviation); unit: number of app uses
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 72 | 80
number of app uses | 40.24 (78.98) | 39.74 (70.22)

30. Primary Outcome: Ease of Use
Description: how easy app was to use (range = 1-7 with higher being easier to use)
Time Frame: 3 weeks (i.e., immediately post-intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 71 | 79
units on a scale | 6.13 (1.19) | 6.27 (1.07)

31. Secondary Outcome: Five Facet Mindfulness Questionnaire Observing Subscale
Description: trait mindfulness observing (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 72 | 80
score on a scale | 22.28 (6.23) | 21.38 (6.2)

32. Secondary Outcome: Five Facet Mindfulness Questionnaire Observing Subscale
Description: trait mindfulness observing (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: 3 weeks (i.e., immediately post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 71 | 79
score on a scale | 22.66 (6.39) | 22.05 (6.22)

33. Secondary Outcome: Five Facet Mindfulness Questionnaire Observing Subscale
Description: trait mindfulness observing (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: 6 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 66 | 76
score on a scale | 23.05 (5.69) | 21.97 (5.74)

34. Secondary Outcome: Five Facet Mindfulness Questionnaire Observing Subscale
Description: trait mindfulness observing (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 64 | 74
score on a scale | 23.77 (5.83) | 22.45 (5.95)

35. Secondary Outcome: Five Facet Mindfulness Questionnaire Observing Subscale
Description: trait mindfulness observing (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: 6 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 63 | 71
score on a scale | 24.19 (5.76) | 21.48 (6.99)

36. Secondary Outcome: Five Facet Mindfulness Questionnaire Describing Subscale
Description: trait mindfulness describing (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 72 | 80
score on a scale | 24.26 (5.75) | 24.69 (5.75)

37. Secondary Outcome: Five Facet Mindfulness Questionnaire Describing Subscale
Description: trait mindfulness describing (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: 3 weeks (i.e., immediately post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 71 | 79
score on a scale | 25 (5.98) | 23.94 (5.1)

38. Secondary Outcome: Five Facet Mindfulness Questionnaire Describing Subscale
Description: trait mindfulness describing (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: 6 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 66 | 76
score on a scale | 25.17 (6.17) | 25.25 (5.35)

39. Secondary Outcome: Five Facet Mindfulness Questionnaire Describing Subscale
Description: trait mindfulness describing (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 64 | 74
score on a scale | 25.55 (5.96) | 24.3 (5.41)

40. Secondary Outcome: Five Facet Mindfulness Questionnaire Describing Subscale
Description: trait mindfulness describing (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: 6 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 63 | 71
score on a scale | 25.56 (6.16) | 24.97 (5.54)

41. Secondary Outcome: Five Facet Mindfulness Questionnaire Awareness Subscale
Description: trait mindfulness acting with awareness (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 72 | 80
score on a scale | 25.03 (6.23) | 26.18 (5.84)

42. Secondary Outcome: Five Facet Mindfulness Questionnaire Awareness Subscale
Description: trait mindfulness acting with awareness (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: 3 weeks (i.e., immediately post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 71 | 79
score on a scale | 25.42 (6.55) | 24.94 (6.41)

43. Secondary Outcome: Five Facet Mindfulness Questionnaire Awareness Subscale
Description: trait mindfulness acting with awareness (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: 6 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 66 | 76
score on a scale | 25.12 (6.34) | 25.7 (5.42)

44. Secondary Outcome: Five Facet Mindfulness Questionnaire Awareness Subscale
Description: trait mindfulness acting with awareness (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 64 | 74
score on a scale | 24.98 (5.9) | 25.27 (5.62)

45. Secondary Outcome: Five Facet Mindfulness Questionnaire Awareness Subscale
Description: trait mindfulness acting with awareness (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: 6 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 63 | 71
score on a scale | 25.43 (6.25) | 26.07 (6.32)

46. Secondary Outcome: Five Facet Mindfulness Questionnaire Nonjudging Subscale
Description: trait mindfulness non-judging of inner experience (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 72 | 80
score on a scale | 25.56 (7.46) | 27.49 (7.58)

47. Secondary Outcome: Five Facet Mindfulness Questionnaire Nonjudging Subscale
Description: trait mindfulness non-judging of inner experience (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: 3 weeks (i.e., immediately post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 71 | 79
score on a scale | 27.86 (6.79) | 27.05 (7.52)

48. Secondary Outcome: Five Facet Mindfulness Questionnaire Nonjudging Subscale
Description: trait mindfulness non-judging of inner experience (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: 6 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 66 | 76
score on a scale | 28.23 (7.23) | 27.93 (6.94)

49. Secondary Outcome: Five Facet Mindfulness Questionnaire Nonjudging Subscale
Description: trait mindfulness non-judging of inner experience (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: 12 weeks post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 64 | 74
score on a scale | 27.88 (7.4) | 27.74 (7.15)

50. Secondary Outcome: Five Facet Mindfulness Questionnaire Nonjudging Subscale
Description: trait mindfulness non-judging of inner experience (range = 8-40 with higher scores indicating greater mindfulness)
Time Frame: 6 months post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 63 | 71
score on a scale | 28.87 (7.45) | 28.01 (6.72)

51. Secondary Outcome: Five Facet Mindfulness Questionnaire Nonreactivity Subscale
Description: trait mindfulness non-reactivity to inner experience (range = 7-35 with higher scores indicating greater mindfulness)
Time Frame: baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 72 | 80
score on a scale | 19.58 (4.58) | 19.44 (3.99)

52. Secondary Outcome: Five Facet Mindfulness Questionnaire Nonreactivity Subscale
Description: trait mindfulness non-reactivity to inner experience (range = 7-35 with higher scores indicating greater mindfulness)
Time Frame: 3 weeks (i.e., immediately post-intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 71 | 79
score on a scale | 20.09 (4.64) | 19.72 (4.34)

53. Secondary Outcome: Five Facet Mindfulness Questionnaire Nonreactivity Subscale
Description: trait mindfulness non-reactivity to inner experience (range = 7-35 with higher scores indicating greater mindfulness)
Time Frame: 6 weeks post intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 66 | 76
score on a scale | 20.72 (5.61) | 19.65 (4.26)

54. Secondary Outcome: Five Facet Mindfulness Questionnaire Nonreactivity Subscale
Description: trait mindfulness non-reactivity to inner experience (range = 7-35 with higher scores indicating greater mindfulness)
Time Frame: 12 weeks post intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 64 | 74
score on a scale | 21.19 (4.16) | 20.14 (3.86)

55. Secondary Outcome: Five Facet Mindfulness Questionnaire Nonreactivity Subscale
Description: trait mindfulness non-reactivity to inner experience (range = 7-35 with higher scores indicating greater mindfulness)
Time Frame: 6 months post intervention)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 63 | 71
score on a scale | 21.3 (4.67) | 20.03 (4.52)

56. Secondary Outcome: State Mindfulness Bodily Sensations
Description: average focus on bodily sensations during intervention period rated on visual analog scale (range = 0-100 with higher scores indicating more mindfulness)
Time Frame: 3 weeks (i.e., immediately post-intervention)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 72 | 80
units on a scale | 36.59 (21.06) | 38.67 (21.35)

57. Secondary Outcome: State Mindfulness Present Focus
Description: average % focus on present moment (as opposed to past or future focus) during intervention period indicating more mindfulness
Time Frame: 3 weeks (i.e., immediately post-intervention)
Measure: Mean (Standard Deviation); unit: percentage of time focused on present
Arm/Group | Mindfulness App | Control Condition
Number analyzed (Participants) | 72 | 80
percentage of time focused on present | .633 (.22) | .558 (.23)

ADVERSE EVENTS:
Time Frame: Baseline through 6-month follow-up.
Arm/Group | Mindfulness App | Control Condition
All-Cause Mortality (participants affected / at risk) | 0/72 | 0/80
Serious Adverse Events (participants affected / at risk) | 1/72 | 0/80
Other Adverse Events (participants affected / at risk) | 8/72 | 5/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness App (N=72) | Control Condition (N=80)
Suicide Attempt (Social circumstances) | 1 (1) | 0 (0) — An adolescent participant reported a suicide attempt on their survey. We immediately intervened with both the parent and child. This adolescent was already seeing a mental health professional.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness App (N=72) | Control Condition (N=80)
Stress from noticing negative emotions (Psychiatric disorders) | 1 (1) | 3 (3) — Adolescents rated how anxious or sad they were feeling in the present moment when using the app. Some adolescents reported discomfort surrounding the acknowledgment of negative emotions.
Onset of Non-suicidal Self-Injury (Psychiatric disorders) | 2 (2) | 1 (1) — Adolescents reported the onset of self-injury.
Onset of Passive Suicidal Ideation (Psychiatric disorders) | 3 (3) | 1 (1)
Discomfort from Mindfulness Activity (Psychiatric disorders) | 2 (2) | 0 (0) — One adolescent reported focusing on sounds sometimes made them stressed when they were meditating in a chaotic environment. Another participant noticed that they had a headache once when completing a mindfulness exercise from focusing.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/16/NCT03900416/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/16/NCT03900416/ICF_001.pdf